CLINICAL TRIAL: NCT02384057
Title: Cognitive Rehabilitation for Participants With Stroke or Brain Injury Using C8 Sciences
Brief Title: Cognitive Rehabilitation With C8 Sciences
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Rehabilitation Center, Seoul, Korea (Other Government)
Collaborators: Hanyang University (Other); National IT Industry Promotion Agency, Republic of Korea (Unknown)
Responsible Party: Principal Investigator, Joon-Ho Shin, Team manager, National Rehabilitation Center, Seoul, Korea
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NRC-2013-04-036
Record Dates: First submitted 2015-02-23; First posted 2015-03-10 (Estimated); Last update posted 2018-03-06 (Actual); Status verified 2018-03

CONDITIONS: Stroke; Brain Injuries
MeSH Terms: conditions — Stroke; Brain Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- C8 sciences (Experimental): cognitive rehabilitation with C8 sciences
  Interventions: Other: Computerized cognitive training program
- Conventional cognitive rehabilitation (Active Comparator): cognitive rehabilitation with conventional methods
  Interventions: Other: Conventional cognitive rehabilitation

INTERVENTIONS:
Other: Computerized cognitive training program — 1000 minutes of computerized cognitive rehabilitation with C8 sciences program
  Arms: C8 sciences
Other: Conventional cognitive rehabilitation — Same amount of conventional cognitive rehabilitation
  Arms: Conventional cognitive rehabilitation

SUMMARY:
C8 sciences program is a cognitive training program mainly developed for the students, and the effectiveness is well established. The aim of this trial is to assess clinical efficacy of the program for cognitive rehabilitation of the patients with stroke or brain injury.

ELIGIBILITY:
Inclusion Criteria:

* Participants with stroke or brain injury
* Cognitive deficits

Exclusion Criteria:

* Uncontrolled medical comorbidities
* Not able to perform outcome measurements
* Aphasia, which hamper communication
* Pre-diagnosed psychological or other neurological disease not relevant to stroke or brain injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2014-12; Primary Completion 2017-10-27 (Actual); Study Completion 2017-10-27 (Actual)

PRIMARY OUTCOMES:
Change from baseline Cambridge Neuropsychological Test Automated Battery(CANTAB) Spatial working memory at 34 th intervention | Baseline, 34th day from baseline
Change from baseline CANTAB Rapid Visual information Processing at 34 th intervention | Baseline, 34th day from baseline

SECONDARY OUTCOMES:
CANTAB Spatial working memory | Baseline, 34th day from baseline, 64th day from baseline
CANTAB Rapid Visual information Processing | Baseline, 34th day from baseline, 64th day from baseline
CANTAB Motor control task | Baseline, 34th day from baseline, 64th day from baseline
CANTAB Paired Associated Learning | Baseline, 34th day from baseline, 64th day from baseline
CANTAB reaction time | Baseline, 34th day from baseline, 64th day from baseline
CANTAB Attention Switching Task | Baseline, 34th day from baseline, 64th day from baseline
CANTAB Stoking of Cambridge | Baseline, 34th day from baseline, 64th day from baseline
CANTAB Emotion Recognition Task | Baseline, 34th day from baseline, 64th day from baseline
CANTAB Stop Signal Task | Baseline, 34th day from baseline, 64th day from baseline
Geriatric depression scale | Baseline, 34th day from baseline
  Older participants
Beck depression index | Baseline, 34th day from baseline
Korean Mini-Mental State Examination (K-MMSE) | Baseline, 34th day from baseline
Korean activities of daily living (K-ADL) | Baseline, 34th day from baseline, 64th day from baseline
Korean instrumental activities of daily living (K-IADL) | Baseline, 34th day from baseline, 64th day from baseline
clinical dementia rating scale (CDR) | Baseline, 34th day from baseline
Stroke impact scale | Baseline, 34th day from baseline
Subjective memory complaint questionnaire | Baseline, 34th day from baseline, 64th day from baseline
NIH toolbox | Baseline, 17th day from baseline, 34th day from baseline, 64th day from baseline
Autobiographical memory | Baseline, 34th day from baseline
Trail making test (A/B) | Baseline, 34th day from baseline, 64th day from baseline
Trail making test - Black and White | Baseline, 34th day from baseline, 64th day from baseline

CONTACTS AND LOCATIONS:
Locations (1):
- National Rehabilitation Center, Seoul, South Korea

REFERENCES:
- [Derived] Gibson E, Koh CL, Eames S, Bennett S, Scott AM, Hoffmann TC. Occupational therapy for cognitive impairment in stroke patients. Cochrane Database Syst Rev. 2022 Mar 29;3(3):CD006430. doi: 10.1002/14651858.CD006430.pub3. PMID 35349186